CLINICAL TRIAL: NCT04080245
Title: Functional Consequences of T-bet Expression in Flu-specific Memory B Cells After Live Attenuated Influenza Vaccine (LAIV)
Acronym: LAIV
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Anoma Nellore, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-300003669
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Influenza, Human
Keywords: Vaccine; Influenza; Efficacy
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Group (Experimental)
  Interventions: Biological: Treatment Group Live Attenuated Flu Vaccine (LAIV)

INTERVENTIONS:
Biological: Treatment Group Live Attenuated Flu Vaccine (LAIV) — We will administer LAIV once as a vaccine prime and IIV once as a vaccine boost with serial weekly blood draws for a month to validate a biomarker of LAIV efficacy.

SUMMARY:
As yet the investigators do not understand if there are biomarkers of immune protection after the Flumist or Live Attenuated Flu Vaccine (LAIV). Here the investigators test the hypothesis that the T-bet expressing fraction of flu-specific B cells after live attenuated influenza vaccination also serves as an early biomarker of long-lived antibody responses after vaccination. In this study the investigators will be providing the LAIV to up to 10 healthy subjects and assaying their immune response and then providing the intramuscular influenza vaccination and testing to see if the immune protection after the LAIV also protects after the intramuscular influenza vaccination.

Update: We have amended this protocol to study the antigen-specific B cell populations that circulate after LAIV or IIV prime and LAIV or IIV boost.

DETAILED DESCRIPTION:
Previously (1) the investigators established that a fluorochrome labeled reagent with the influenza antigen hemagglutinin accurately identified flu-specific B cells after inactivated influenza vaccination and we established that a subset of these flu-specfiic B cells that express the lineage defining master transcriptional regulator, T-bet, correlate with long lived antibody responses. As yet the investigators do not understand if there are biomarkers of immune protection after the Flumist or Live Attenuated Flu Vaccine (LAIV). Here the investigators test the hypothesis that the T-bet expressing fraction of flu-specific B cells after live attenuated influenza vaccination also serves as an early biomarker of long-lived antibody responses after vaccination. In this study the investigators will be providing the LAIV to up to 10 healthy subjects and assaying their immune response and then providing the intramuscular influenza vaccination and testing to see if the immune protection after the LAIV also protects after the intramuscular influenza vaccination.

Update: We have amended this protocol to study the antigen-specific B cell populations that circulate after LAIV or IIV prime and LAIV or IIV boost.

ELIGIBILITY:
Inclusion Criteria:

* Missed getting the flu vaccine in the last year
* No history of reactive airway disease
* No history of allergy to LAIV
* No history of allergy to IIV
* Self-identify as healthy without an immunocompromising condition defined as cancer, autoimmune disease, organ transplant or receipt of steroids.

Exclusion Criteria:

* History of reactive airway disease
* History of allergy to LAIV or IIV
* Do not self-identify as healthy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Outcome Measure: Participants with a positive T-bet expressing Flu-specific B cell subtype | Baseline
  The investigators will perform a blood test on lymphocytes from circulating blood.
Outcome Measure: Participants with a positive T-bet expressing Flu-specific B cell subtype | 7 days post first injection
  The investigators will perform a blood test on lymphocytes from circulating blood.
Outcome Measure: Participants with a positive T-bet expressing Flu-specific B cell subtype | 14 days post first injection
  The investigators will perform a blood test on lymphocytes from circulating blood.
Outcome Measure: Participants with a positive T-bet expressing Flu-specific B cell subtype | 7 days post second injection
  The investigators will perform a blood test on lymphocytes from circulating blood.

CONTACTS AND LOCATIONS:
Overall Officials: Anoma Nellore, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No